CLINICAL TRIAL: NCT02542423
Title: Endocan Predictive Value in Postcardiac Surgery Acute Respiratory Failure. The ENDOLUNG Study
Brief Title: Endocan Predictive Value in Postcardiac Surgery Acute Respiratory Failure.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Principal Investigator, Andrea PERROTTI, Medical Doctor, Centre Hospitalier Universitaire de Besancon
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CPP 15/479
Record Dates: First submitted 2015-09-01; First posted 2015-09-07 (Estimated); Last update posted 2015-09-07 (Estimated); Status verified 2015-09

CONDITIONS: Respiratory Failure; Postoperative Complications
MeSH Terms: conditions — Respiratory Insufficiency; Postoperative Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- patients undergoing cardiac surgery (Other)
  Interventions: Other: Endocan blood test samples

INTERVENTIONS:
Other: Endocan blood test samples
  Other Names: Endocan; Endolung

SUMMARY:
According to literature data, Endocan can detect the onset of respiratory failure. The investigators aim to prove its value also for cardiac surgery patients.

DETAILED DESCRIPTION:
Endocan is an endothelium derived soluble dermatan sulfate proteoglycan. Literature data shows that alterate levels of its blood concentration correlate with the onset of pulmonary failure in patients with major trauma and septic shock.

In cardiac surgery respiratory failure and infections are threatening complications leading to mortality rates up to 80%. A rapid diagnosis and treatment of this pathology is crucial to improve the clinical outcome.

Unfortunately specific data for the efficacy of Endocan predictive value in cardiac surgery patients are not available.

The investigators aim to determinate if Endocan can be a helpful tool to identify patients developing acute respiratory failure after cardiac surgery and anticipate specific treatment in order to improve survival.

ELIGIBILITY:
Inclusion Criteria:

* Able to give written consent
* Elective cardiac surgery
* More than 18 years old

Exclusion Criteria:

* Less than 18 years old
* urgency / emergency cardiac surgery
* pregnancy
* refusal
* unable to give written consent
* oncologic patients
* concomitant inflammatory or infective pulmonary disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2015-09; Primary Completion 2016-03 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Changes of Endocan blood levels after cardiac surgery and its correlation with postoperative pulmonary failure | from day -1 of the intervention to day 3, one blood sample per day
  The investigators will enroll 150 patients undergoing elective cardiac surgery. Every participant will be prelevated of several blood samples following this time frame : day -1 from intervention, day 0 ( six hours after intervention), day 1 , day 2 , day 3. All patients will be observed to detect all infections, especially pulmonary ones, up to hospital discharge. Endocan blood levels of patients developing pulmonary failure and patients without postoperative respiratory insufficiency will be compared.

REFERENCES:
- [Derived] Chazal E, Morin L, Chocron S, Lassalle P, Pili-Floury S, Salomon du Mont L, Ferreira D, Samain E, Perrotti A, Besch G. Impact of early postoperative blood glucose variability on serum endocan level in cardiac surgery patients: a sub study of the ENDOLUNG observational study. Cardiovasc Diabetol. 2023 Aug 24;22(1):221. doi: 10.1186/s12933-023-01959-5. PMID 37620974